CLINICAL TRIAL: NCT05289739
Title: Get Strong to Fight Childhood Cancer: An Exercise Intervention for Children and Adolescents Undergoing Anti-Cancer Treatment
Brief Title: Exercise Training in Childhood Cancer
Acronym: FORTEe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: University Hospital Heidelberg (Other); Centre Leon Berard (Other); Oxford Brookes University (Other); Fondazione Monza e Brianza per il Bambino e la sua Mamma (MBBM) (Other); European University of Madrid (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); University Medical Centre Ljubljana (Other); Rigshospitalet, Denmark (Other); German Sport University, Cologne (Other); University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Joerg Faber, Univ. Prof. Dr. med., Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMC-Mainz: 21-00338
Record Dates: First submitted 2022-01-18; First posted 2022-03-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pediatric Oncology
Keywords: Paediatric exercise oncology; precision exercise training; childhood cancer; randomized controlled trial; quality of life; augmented reality; exercise technology
MeSH Terms: conditions — Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Usual medical care + supervised exercise training during intensive medical treatment
  Interventions: Behavioral: Exercise training
- Control group (No Intervention): Usual medical care

INTERVENTIONS:
Behavioral: Exercise training — Exercise training during intensive cancer treatment. Training mainly consists of age-appropriate and personalized endurance, strength, flexibility, balance/coordination and gait training. Three to five weekly training sessions lasting 30 to 60 minutes each for about eight to ten weeks (depending on the course of the cancer treatment).
  Arms: Exercise group

SUMMARY:
The purpose of this multicenter study is to evaluate a personalised and standardised exercise intervention for children and adolescents undergoing anti-cancer treatment.

DETAILED DESCRIPTION:
In the randomised, controlled FORTEe trial, high evidence for an innovative, patient-centred exercise treatment shall be generated. Supervised exercise training intents to increase muscle strength and reduce muscular atrophy due to bedrest. CRF and HRQoL can be improved and in the future, these benefits may help to fight childhood cancer by increasing therapy efficiency and survival rate. Within the project, digital, innovative technologies such as augmented reality will be developed and applied to make the exercise training more effective, age-adapted and personalised. Moreover, FORTEe will stimulate translational research to provide access to paediatric exercise oncology as a new health care intervention. As a progress beyond the current state-of-the-art, FORTEe has the ambition to implement paediatric exercise oncology as an evidence-based standard in clinical care for all childhood cancer patients across the EU and beyond.

ELIGIBILITY:
Inclusion criteria:

* First/initial diagnosis of a primary oncologic disease according to the International Classification of Childhood Cancer (ICCC), requiring chemotherapy and/or radiation therapy or First/initial diagnosis of a relapsed oncologic disease according to the International Classification of Childhood Cancer (ICCC), requiring chemotherapy and/or radiation therapy or First/initial diagnosis of a secondary oncologic disease according to the International Classification of Childhood Cancer (ICCC), requiring chemotherapy and/or radiation therapy
* Planned or started anti-cancer treatment (chemo- and/or radiotherapy) at one of the recruiting centres of the FORTEe trial
* The patient is assessed by the treating team (pediatric oncologist, exercise professional etc.) as suitable to participate in the trial, e.g. due to medical or psychological reasons.
* Existing informed consent (or assent) to participate in the study
* The patient (and the legal guardian) has/have sufficient knowledge of the respective national or English language so that it is possible to carry out the informed consent as well as interviews (in age-appropriate language).
* The patient is not in a terminal phase of the disease.

Exclusion criteria:

* Oncologic disease (primary/relapsed/secondary) according to the International Classification of Childhood Cancer (ICCC), requiring neither chemotherapy nor radiation therapy or solely requiring surgery
* Reasons that already exist or are foreseeable at the time of study enrolment, due to which the patient will not have access to the exercise intervention and/or to the pre-test and/or to the post-test (e.g. foreseeable or planned, permanent change of treatment centre)
* The patient is assessed by the treating team (pediatric oncologist, exercise professional etc.) as unsuitable to participate in the trial, e.g. due to medical or psychological reasons.
* After detailed information and, if necessary, having time to consider, the patient (≥ 16 years of age) did not agree to give written informed consent to participate in the trial.
* The patient (and the legal guardians) has/have insufficient knowledge of the respective national or English language, so that it is not possible to carry out both the informed consent and interviews (in age-appropriate language).
* The patient is in a terminal phase of the disease

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 478 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2026-01-26 (Actual); Study Completion 2026-01-26 (Actual)

PRIMARY OUTCOMES:
Change in the score of Cancer-related fatigue during the intervention, after the intervention, and over a 1-year follow-up period compared with baseline | pre-intervention; bi-weekly during the intervention (up to 10 weeks); end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention; after intensive cancer treatment; 15 months after the end of intervention
  Cancer-related fatigue measured by the Pediatric Quality of Life Inventory (PedsQL) 3.0 Multidimensional Fatigue Scale. The PedsQL Multidimensional Fatigue Scale is composed of 18 items comprising three dimensions. Scores are transformed on a scale from 0 to 100. Higher scores indicate lower fatigue.

SECONDARY OUTCOMES:
Change in the score of general Health-Related Quality of Life during the intervention, after the intervention, and over a 1-year follow-up period compared with baseline | pre-intervention; bi-weekly during the intervention (up to 10 weeks); end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention; after intensive cancer treatment; 15 months after the end of intervention
  Health-Related Quality of Life measured by the Measurement Model for the Pediatric Quality of Life Inventory (PedsQL) 4.0 Generic Core Scales questionnaire.
  On the PedsQL Generic Core Scales, for ease of interpretability, items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL (Health-Related Quality of Life).
Change in the score of cancer-related Health-Related Quality of Life during the intervention, after the intervention, and over a 1-year follow-up period compared with baseline | pre-intervention; bi-weekly during the intervention (up to 10 weeks); end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention; after intensive cancer treatment; 15 months after the end of intervention
  Health-Related Quality of Life measured by the Measurement Model for the Pediatric Quality of Life Inventory (PedsQL) 3.0 Cancer Module questionnaire.
  Scores are transformed to a 0 to 100 scale. Higher scores indicate lower problems.
Change in the score of Mental Health (measured by WHO (Five) Well-Being Index) during the intervention, after the intervention, and over a 1-year follow-up period compared with baseline | pre-intervention; bi-weekly during the intervention (up to 10 weeks); end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention; after intensive cancer treatment; 15 months after the end of intervention
  WHO (Five) Well-Being Index (1998 version) is used to measure Mental Health.The WHO-5 consists of five statements, which respondents rate according to the scale below:
  All of the time = 5 Most of the time = 4 More than half of the time = 3 Less than half of the time = 2 Some of the time = 1 At no time = 0. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Change in the score of Mental Health (measured by Warwick-Edinburgh Mental Well-being Scale (WEMWBS)) during the intervention, after the intervention, and over a 1-year follow-up period compared with baseline | pre-intervention; bi-weekly during the intervention (up to 10 weeks); end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention; after intensive cancer treatment; 15 months after the end of intervention
  Warwick-Edinburgh Mental Well-being Scale (WEMWBS) is used to measure Mental Health. WEMWBS is a 14 item scale of mental well-being covering subjective well-being and psychological functioning, in which all items are worded positively and address aspects of positive mental health. The total score of the 14-item scale WEMWBS is obtained by summing the score for each of the 14 items. The scoring range for each item is from 1 - 5 and the total score is from 14-70.
Change in the score of Resilience (measured by Mainzer Resilience Scale for childhood cancer (MRScc)) during the intervention, after the intervention, and over a 1-year follow-up period compared with baseline | pre-intervention; bi-weekly during the intervention (up to 10 weeks); end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention; after intensive cancer treatment; 15 months after the end of intervention
  Stress reactivity measured by the Mainz Resilience Score for childhood cancer (MRScc). The MRScc consists of 4 dimensions on mental health problems and 6 dimensions on stressor exposure. For both categories mental health problems and stressor exposure 4 - 400 points can be achieved. To calculate the resilience score, the category mental health problems is divided by the category stressor exposure. A score >0 means low resilience, a score < 0 means high resilience.
Change in the score of Resilience (measured by the Brief Resilience Scale (BRS)) during the intervention, after the intervention, and over a 1-year follow-up period compared with baseline | pre-intervention; bi-weekly during the intervention (up to 10 weeks); end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention; after intensive cancer treatment; 15 months after the end of intervention
  Resilience will be evaluated using the Brief Resilience Scale (BRS). BRS is a 6 item scale, the items are rated from 1 to 5. A total score is calculated by determining the sum of the individual items which result in a total score ranging from 6 to 30. A higher score means a higher resilience.
Change in the score of Resilience (measured by the Child & Youth Resilience Measure-Revised (CYRM-R)) during the intervention, after the intervention, and over a 1-year follow-up period compared with baseline | pre-intervention; bi-weekly during the intervention (up to 10 weeks); end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention; after intensive cancer treatment; 15 months after the end of intervention
  Resilience will be evaluated using the Child & Youth Resilience Measure-Revised (CYRM-R).
  The items within the measures can be directly summed to gain a total score of an individual's resilience. For the unmodified 5-point measure (with responses going from 1-5), the minimum score is 17 and the maximum score is 85. For the overall measure and subscales, higher scores indicate characteristics associated with resilience.
Change in the score of General self-efficacy during the intervention, after the intervention, and over a 1-year follow-up period compared with baseline | pre-intervention; bi-weekly during the intervention (up to 10 weeks); end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention; after intensive cancer treatment; 15 months after the end of intervention
  General self-efficacy will be evaluated using the General self-efficacy scale (GSE). The total score is calculated by finding the sum of the 10 items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Change in the score of Physical exercise self-efficacy during the intervention, after the intervention, and over a 1-year follow-up period compared with baseline | pre-intervention; bi-weekly during the intervention (up to 10 weeks); end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention; after intensive cancer treatment; 15 months after the end of intervention
  Physical self-efficacy will be evaluated using the Physical exercise self-efficacy scale (PESE). The total score is calculated by finding the sum of the 10 items. For the GSE, the total score ranges between 5 and 20, with a higher score indicating more self-efficacy.
Change in the Physical activity level (measured by the Modifed Recent Physical Activity Questionnaire (mRPAQ)) during the intervention, after the intervention, and over a 1-year follow-up period compared with baseline | pre-intervention; bi-weekly during the intervention (up to 10 weeks); end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention; after intensive cancer treatment; 15 months after the end of intervention
  Physical activity level will be evaluated using the Modifed Recent Physical Activity Questionnaire (mRPAQ).
  The duration of listed physical activities were reported (recall time: over the past 7 days). Descriptive Statistics will be performed.
Change in the Physical activity level (measured by the Modified Youth Physical Activity Questionnaire (mYPAQ)) during the intervention, after the intervention, and over a 1-year follow-up period compared with baseline | pre-intervention; bi-weekly during the intervention (up to 10 weeks); end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention; after intensive cancer treatment; 15 months after the end of intervention
  Physical activity level will be evaluated using Modified Youth Physical Activity Questionnaire (mYPAQ).
  The duration of listed physical activities were reported (recall time: over the past 7 days). Descriptive Statistics will be performed.
Change in the Physical activity level (measured by the Modified Children's Physical Activity Questionnaire (mCPAQ)) during the intervention, after the intervention, and over a 1-year follow-up period compared with baseline | pre-intervention; bi-weekly during the intervention (up to 10 weeks); end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention; after intensive cancer treatment; 15 months after the end of intervention
  Physical activity level will be evaluated using Modified Children's Physical Activity Questionnaire (mCPAQ).
  The duration of listed physical activities were reported (recall time: over the past 7 days). Descriptive Statistics will be performed.
Change in the Physical activity level and behaviour during the intervention, after the intervention, and over a 1-year follow-up period compared with baseline | pre-intervention; bi-weekly during the intervention (up to 10 weeks); end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention; after intensive cancer treatment; 15 months after the end of intervention
  In a semi-structured interview on physical activity, qualitative data will be collected regarding activity behaviour, motivating factors and barriers to physical activity.
Change in functional capacity after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  Measured via Six Minute Walk Test (6MWT). Functional capacity is evalauted by the walked distance.
Change in endurance performance (measured by the assisted 6-minute cycling test) after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  Measured via assisted 6-minute cycling test (A6MCT). Endurance performance is evaluated by the cumulative revolutions after 6 minutes.
Change in endurance performance (measured by the adapted Yo-Yo-Test) after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  Endurance performance will be evaluated by the adapted Yo-Yo-Test.
Longitudinal assessment of oxidative skeletal muscle impairment after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  Muscle impairment will be evaluated by near infrared spectroscopy (NIRS).
Change in peak oxygen uptake (VO2peak) after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  Cardiopulmonary Exercise Testing (CPET) will be performed during an endurance test to exhaustion to determine the peak oxygen uptake (VO2peak).
Change in motor function after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  measured via the quick motor function test
Change in hamstrings flexibility after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  measured via the sit and reach test
Change in lower limbs flexibility after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  a goniometer is used to measure the angles during foot, knee and hip flexion
Change in functional strength after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  Functional strength will be evaluated using the sit to stand test.
Change in arm strength after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  Arm strength will be evaluated using 5 repetition maximum for biceps curls.
Change in upper body strength after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  Upper body strength will be evaluated using medicine ball shot test.
Change in knee flexor strength after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  Knee flexor strength will be evaluated using a handheld dynamometer.
Change in leg extension strength after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  Leg extension strength will be evaluated using 5 repetition maximum for leg extension test measured via leg extension machine.
Change in functional mobility after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  Functional mobility will be evaluated using the timed up and down stairs test (TUDS).
Change in static balance after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  Static balance will be determined with the static stand test.
Change in body composition (measured via skinfold measurement) after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  Body composition is measured via plicometry of the triceps.
Change of the phase angle by means of bioelectrical impedance analysis for the examination of body composition after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  A multifrequency (5, 50, 100 kHz) bioelectrical impedance analysis is performed using a phase-sensitive impedance analyser (BIAcorpus RX4004M). For this purpose, a sinusoidal alternating current with a constant intensity is applied to the patient's wrists and ankles. The phase angle (PA, ° degree) is measured by the impedance analyser as the phase shift between current and voltage. The phase angle provides conclusions about nutritional status and body composition.
Change in body composition (measured via dual-energy x-ray absorptiometry) after the intervention and after a 12-week follow-up compared to baseline | pre-intervention; end of intervention (assessed up to 10 weeks); 12 weeks after the end of intervention
  In the dual energy X-ray absorptiometry (DEXA) total muscle mass and total fat mass is determined.
Usage frequency of the augmented reality (AR) app from baseline to the end of app use | during the use of the app from baseline until the end of app use (15 months after the end of intervention)
  Usage frequency derived from dates within an exercise diary is recorded during the entire time the AR (augmented reality) app is used.
Usability of the augmented reality app | post app use (15 months after the end of intervention)
  Exploration of app usability via user experience, incl. functions/features, technical bugs. For this purpose, qualitative data will be collected in a semi-structured interview.
Usability of the pixformance station | post app use (15 months after the end of intervention)
  The pixformance station is a digital training tool. Pixformance usability should be explored through user experience, incl. functions/features, and technical bugs. For this purpose, qualitative data will be collected in a semi-structured interview.
Composite multidimensional socioeconomic status index | pre-intervention
  Socioeconomic status will be assessed in order to perform a confounder analysis for the main outcome cancer-related fatigue.
  The calculation of the socioeconomic status index is based on the dimensions "levels of education", "occupational status" and "income". Scores for each dimension ranged from 1 to a maximum of 7. Since the 3 subscales are included in the calculation with the same weight, the socioeconomic status index can assume values between 3.0 and 21.0. Higher scores mean higher socioeconomic status.
Change in the number of T-cells before start of anti-cancer treatment (baseline), pre-exercise intervention and post-exercise intervention | Blood sampling before start of anti-cancer treatment (chemo- and/or radiotherapy); pre-intervention; end of intervention (assessed up to 10 weeks)
  The purpose of the biomarker analysis is to describe peripheral circulating immune cell profiles and DNA methylation status at baseline (T-1) (i.e. before chemo- and/or radiotherapy), and pre- (T0) and post-exercise intervention (T1) (both during chemo- and/or radiotherapy) solely in adolescent and young adult patients suffering from a solid tumour excluding cancers of the immune system e.g. leukemia and lymphoma.
Change in the number of B-cells before start of anti-cancer treatment (baseline), pre-exercise intervention and post-exercise intervention | Blood sampling before start of anti-cancer treatment (chemo- and/or radiotherapy); pre-intervention; end of intervention (assessed up to 10 weeks)
  The purpose of the biomarker analysis is to describe peripheral circulating immune cell profiles and DNA methylation status at baseline (T-1) (i.e. before chemo- and/or radiotherapy), and pre- (T0) and post-exercise intervention (T1) (both during chemo- and/or radiotherapy) solely in adolescent and young adult patients suffering from a solid tumour excluding cancers of the immune system e.g. leukemia and lymphoma.
Change in the number of NK-cells before start of anti-cancer treatment (baseline), pre-exercise intervention and post-exercise intervention | Blood sampling before start of anti-cancer treatment (chemo- and/or radiotherapy); pre-intervention; end of intervention (assessed up to 10 weeks)
  The purpose of the biomarker analysis is to describe peripheral circulating immune cell profiles and DNA methylation status at baseline (T-1) (i.e. before chemo- and/or radiotherapy), and pre- (T0) and post-exercise intervention (T1) (both during chemo- and/or radiotherapy) solely in adolescent and young adult patients suffering from a solid tumour excluding cancers of the immune system e.g. leukemia and lymphoma.
Change in the number of leukocytes before start of anti-cancer treatment (baseline), pre-exercise intervention and post-exercise intervention | Blood sampling before start of anti-cancer treatment (chemo- and/or radiotherapy); pre-intervention; end of intervention (assessed up to 10 weeks)
  The purpose of the biomarker analysis is to describe peripheral circulating immune cell profiles and DNA methylation status at baseline (T-1) (i.e. before chemo- and/or radiotherapy), and pre- (T0) and post-exercise intervention (T1) (both during chemo- and/or radiotherapy) solely in adolescent and young adult patients suffering from a solid tumour excluding cancers of the immune system e.g. leukemia and lymphoma.
Change in the number of monocytes before start of anti-cancer treatment (baseline), pre-exercise intervention and post-exercise intervention | Blood sampling before start of anti-cancer treatment (chemo- and/or radiotherapy); pre-intervention; end of intervention (assessed up to 10 weeks)
  The purpose of the biomarker analysis is to describe peripheral circulating immune cell profiles and DNA methylation status at baseline (T-1) (i.e. before chemo- and/or radiotherapy), and pre- (T0) and post-exercise intervention (T1) (both during chemo- and/or radiotherapy) solely in adolescent and young adult patients suffering from a solid tumour excluding cancers of the immune system e.g. leukemia and lymphoma.
Change in the DNA methylation status of T cells before start of anti-cancer treatment (baseline), pre-exercise intervention and post-exercise intervention | Blood sampling before start of anti-cancer treatment (chemo- and/or radiotherapy); pre-intervention; end of intervention (assessed up to 10 weeks)
  The purpose of the biomarker analysis is to describe peripheral circulating immune cell profiles and DNA methylation status at baseline (T-1) (i.e. before chemo- and/or radiotherapy), and pre- (T0) and post-exercise intervention (T1) (both during chemo- and/or radiotherapy) solely in adolescent and young adult patients suffering from a solid tumour excluding cancers of the immune system e.g. leukemia and lymphoma.
Change in the DNA methylation status of NK cells before start of anti-cancer treatment (baseline), pre-exercise intervention and post-exercise intervention (baseline), pre-exercise intervention and post-exercise intervention | Blood sampling before start of anti-cancer treatment (chemo- and/or radiotherapy); pre-intervention; end of intervention (assessed up to 10 weeks)
  The purpose of the biomarker analysis is to describe peripheral circulating immune cell profiles and DNA methylation status at baseline (T-1) (i.e. before chemo- and/or radiotherapy), and pre- (T0) and post-exercise intervention (T1) (both during chemo- and/or radiotherapy) solely in adolescent and young adult patients suffering from a solid tumour excluding cancers of the immune system e.g. leukemia and lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Faber, Univ.-Prof. Dr. med., Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- Johannes-Gutenberg-University Medical Center, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Derived] Neu MA, Dreismickenbecker E, Lanfranconi F, Stossel S, Balduzzi A, Wright P, Windsor S, Wiskemann J, El-Rajab I, Lucia A, Fiuza-Luces C, Mongondry R, Fridh MK, Spreafico F, Konda B, Kitanovski L, Heisserer B, Polak M, Baader T, Bloch W, Gotte M; Network ActiveOncoKids; Rizvi K; Youth Cancer Europe; Ruckes C, Paul NW, Faber J; FORTEe Consortium. Get strong to fight childhood cancer - an exercise intervention for children and adolescents undergoing anti-cancer treatment (FORTEe): Rationale and design of a randomized controlled exercise trial. BMC Cancer. 2025 Aug 7;25(1):1275. doi: 10.1186/s12885-025-14489-y. PMID 40775303